CLINICAL TRIAL: NCT07361120
Title: Prospective, Multicenter, Single-arm, Open Label, Interventional Clinical Trial Investigating the Safety and Effectiveness of the Plan A Male Contraceptive System.
Brief Title: Plan A Occlusion and Reversal System Feasibility Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Next Life Sciences (Industry)
Collaborators: Clinico Pty Ltd (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CIP102
Record Dates: First submitted 2025-12-16; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Fertility; Fertility, Male; Healthy Male Adults
Keywords: Vasectomy, Fertility, Reproductive Health, Male Contraception, Vas Occlusion, No Scalpel Vasectomy,

STUDY DESIGN:
Intervention Model Description: Group 1 will include 30 subjects that will be followed for up for a maximum of 6 months post occlusion procedure, or until they achieve azoospermia at which point they will be offered a vasectomy procedure. Group 2 will recruit ten subjects who will be followed for up for a maximum of 6 months post occlusion procedure, or until they achieve azoospermia at which point they will have the reversal procedure using the Plan A RD (Reversal Device). This group will be followed for up to another 3 months maximum, or until baseline semen levels are achieved at which point they will be offered a vasectomy procedure. Ten men (all sites) reaching azoospermia after their occlusion procedure will be allocated to Group 2 and will go on to have the reversal procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Occlusion Procedure (Experimental): This will be Group 1. Group1 will have the occlusion procedure but will not have the reversal procedure.
  Interventions: Device: Occlusion System
- Group 2: Reversal Procedure (Experimental): This will be Group 2. Group 2 will have both the occlusion and reversal procedure.
  Interventions: Device: Occlusion System

INTERVENTIONS:
Device: Occlusion System — The occlusion system comprised of the Delivery Lumen Access Device and Vasalgel.

SUMMARY:
Prospective, multicenter, single-arm, open label, interventional clinical trial investigating the safety and effectiveness of the Plan A Male Contraceptive System to occlude the vas deferens to block the passage of sperm and then be reversed to subsequently allow the passage of sperm through the vas deferens.

DETAILED DESCRIPTION:
Prospective, multicenter, single-arm, open label, interventional clinical trial investigating the safety and effectiveness of the Plan A Male Contraceptive System to occlude the vas deferens to block the passage of sperm and then be reversed to subsequently allow the passage of sperm through the vas deferens. 40 men (all sites) will be enrolled and treated with Plan A occlusion (Vasalgel®) using DLAD (Delivery Lumen Access Device). The study will enroll into two groups. Group 1 will include 30 subjects that will be followed for up for a maximum of 6 months post occlusion procedure, or until they achieve azoospermia at which point they will be offered a vasectomy procedure. Group 2 will recruit ten subjects who will be followed for up for a maximum of 6 months post occlusion procedure, or until they achieve azoospermia at which point they will have the reversal procedure using the Plan A RD (Reversal Device). This group will be followed for up to another 3 months maximum, or until baseline semen levels are achieved at which point they will be offered a vasectomy procedure. Ten men reaching azoospermia after their occlusion procedure will be allocated to Group 2 and will go on to have the reversal procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Male subject who is seeking and suitable to undergo a vasectomy as a long-term form of contraception
2. Male subject who has voluntarily signed and dated the Institutional Review Board (IRB)/Ethics Committee (EC) approved informed consent form (ICF) for this study prior to initiation of any screening or study specific procedures
3. 25 to 65 years of age at the time of consent
4. Body Mass Index (BMI) <31 kg/m2
5. Good health for undergoing a vasectomy as confirmed by medical history, physical examination and clinical laboratory tests of blood and urine at the time of screening
6. Normal semen analysis defined by the WHO Laboratory Manual for the Examination and Processing of Human Semen (6th Edition), based on the average of two semen samples ≥2 days and ≤7 days apart
7. In the opinion of the Investigator, subject is suitable to undergo a vasectomy as a form of long-term contraception
8. Agreement to use an effective method of contraception during the entire clinical trial until the planned vasectomy
9. Lives in close proximity to the trial site to enable provision of fresh semen samples unless the subject agrees to provide semen samples at the trial site or laboratory

Exclusion Criteria:

1. (On exam, has any of the following); one or both vasa not present, abnormal scrotum, large varicocele, hydrocele, filariasis or elephantiasis of scrotum, or intrascrotal mass that would make the subject not suitable for the study.
2. Prior testicular surgery, testicular injury or prior vasectomy with vasovasostomy (vasectomy reversal)
3. Recurrent pain with ejaculations
4. Has known allergic reaction to sulfur-containing products or has had a prior severe allergic response to injectable or implantable devices
5. Has local genital infections such as balanitis, scrotal skin infection, epididymitis, or orchitis, or tender (inflamed) tip of the penis, but may be enrolled after resolution of an acute infection
6. History of prostatitis or benign prostatic hypertrophy requiring treatment
7. Has undergone prior chemotherapy
8. Has known current coagulopathy or other bleeding disorders
9. Currently taking or planning to take any type of systemic medication which could affect sperm count or ejaculation (e.g., anabolic steroids, chemotherapy, alpha blocker)
10. Subjects with cystic fibrosis
11. Subjects with a history of inguinal hernia repair
12. Vulnerable subjects (e.g., subjects with cognitive challenges, incarcerated, etc.)
13. Currently participating in another study involving an investigational device or drug (or has participated in a study within the last 30 days prior to screening).
14. Any site staff member with delegated study responsibilities or a family member of a site staff member with delegated study responsibilities
15. In the opinion of the Investigator, there are issues or concerns that may compromise the safety of the subject or confound the reliability of compliance and information acquired in this study
16. Has any condition that, in the opinion of the Investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results.

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Study subjects achieving azoospermia | Starting at the 30 day follow-up visit
  Total number of subjects (N=40) achieving azoospermia
Study subjects that return to baseline semen levels | Correlating to Outcome 1, that follow-up timepoint at which azoospermia is reached starting at the 30 day follow-up
  Total number of subjects (N=10) that return to baseline semen levels after reversal
Adverse Events | From the first subjects screening visit through the last subjects 14 Day phone follow up visit.
  Rate and severity of adverse events.
Subject Comfort | From the first subjects occlusion visit until the last subjects 14 Day phone follow up visit.
  Subject Comfort Assessment Scale Post Occlusion and Reversal
Histology | From the first subjects occlusion visit until the last subjects vasectomy, approximately 9 months
  Excised portion of the vas deferens will be prepared with formalin for histological evaluation

SECONDARY OUTCOMES:
Subject Satisfaction/Comfort Assessment | From the first subjects occlusion visit until the last subjects 14 Day phone follow up visit.
  Patient satisfaction questions along with NRS pain scale are being utilized to determine the comfort of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Homi Zargar, MD, Principal Investigator — Western Urology
Locations (1):
- Western Urology, Maribyrnong, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No